CLINICAL TRIAL: NCT03525405
Title: A Phase I, Open Label, Single Dose Study to Evaluate the Mass Balance of 14C-Napabucasin in Healthy Adult Male Subjects
Brief Title: A Study to Evaluate the Mass Balance of 14C-Napabucasin in Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBI608-104
Record Dates: First submitted 2018-04-30; First posted 2018-05-15 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: ADME; Healthy
MeSH Terms: interventions — napabucasin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Dose (Experimental)
  Interventions: Drug: napabucasin

INTERVENTIONS:
Drug: napabucasin — Single 240 mg dose containing 100 μCi of 14C-napabucasin will be administered with 240 mL of water following an overnight fast.
  Other Names: BBI-608; BBI608

SUMMARY:
This is a Phase I, single-center, open-label, single-sequence, study evaluating the absorption, metabolism, and excretion of napabucasin in healthy adult male volunteers using a mixture 14C-radiolabeled and unlabeled material.

ELIGIBILITY:
Inclusion criteria

1. An Institutional Review Board (IRB) approved informed consent is signed and dated prior to any study-related activities.

2. Subject is male. 3. Subject is between the ages of 18 and 45 years, inclusive at screening. 4. Subject has a body mass index between 18 and 34 kg/m^2 (weight/[height]^2) inclusive at screening.

5. Subject has normal (or abnormal and clinically insignificant according to the Investigator) laboratory values at screening. 6. Subject is in good health, determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs measurements, or clinical laboratory evaluations at Screening or Check-in Day -1 as assessed by the Investigator (or designee). Subject has the ability to understand the requirements of the study and a willingness to comply with all study procedures.

7. Subject has not consumed and agrees to abstain from taking any dietary supplements, herbal products, and non-prescription drugs (except as authorized by the Investigator and Medical Monitor) for 14 days prior to clinical research unit (CRU) admission through follow-up call.

8. Subject has not consumed and agrees to abstain from taking any prescription drugs (except as authorized by the Investigator and Medical Monitor) during the 14 days prior to CRU admission through follow-up call.

9. Subject has not consumed alcohol-containing beverages for 3 days prior to CRU admission and agrees not to consume alcohol through clinic discharge. 10. Subject has not consumed char-broiled meats, cruciferous vegetables, and grapefruit-, apple-, or Seville orange-containing products within the 3 days prior to CRU admission and agrees not to consume Seville oranges, grapefruit and grapefruit juice through clinic discharge.

11. Subject has not used tobacco- and nicotine-containing products within 2 months prior to the CRU admission and agrees to abstain from using tobacco- and nicotine-containing products through clinic discharge.

12. Subject agrees to abstain from consuming caffeine- or xanthine-containing products from 3 days prior to CRU admission through clinic discharge.

13. History of a minimum of 1 bowel movement per day Exclusion criteria

1. Subject has a history of illicit drug abuse in the past year or displays current evidence of such abuse in the opinion of the Investigator.
2. Subject has positive findings on urine drug screen (including cotinine).
3. Subject is positive for human immunodeficiency virus (HIV), hepatitis B and/or hepatitis C on Screening assessments.
4. Subject has a QTcF >450 msec at screening (confirmed by repeat).
5. Subject has a female partner who is either pregnant, nursing, or planning to become pregnant during the study or within 90 days after the last dose of the study drug, or unwilling to follow the contraception requirements.
6. Subject has a clinically significant acute illness within 1 week of CRU admission, or symptoms of active illness at check-in, at discretion of the Investigator (or designee).
7. Subject has a hypersensitivity or allergy to napabucasin or the ingredients of napabucasin, or other clinically significant allergies in the opinion of the Investigator.
8. Subject has donated plasma within 7 days of drug administration.
9. Subject has donated 1 or more pints of blood (or equivalent blood loss) within 30 days prior to drug administration.
10. Subject has a history of chronic Gastroesophageal reflux disease (GERD) or has used omeprazole or other proton pump inhibitors within 3 months of Screening.
11. Subject has congenital non-hemolytic hyperbilirubinemia [e.g., Gilbert's syndrome].
12. Subject has any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy, or other gastrointestinal tract surgery, except appendectomy).
13. Subject has participated in an investigational drug study within 30 days or 5 half-lives (whichever is longer) of exposure to another investigational medication prior to CRU admission.
14. Subject is an employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, or a family member of the employees or the Investigator.
15. Subjects with exposure to significant diagnostic or therapeutic radiation (e.g., serial Xray, computed tomography scan, barium meal) or employment in a job requiring radiation exposure monitoring within 12 months prior to check-in.
16. Subjects who have participated in a radiolabeled drug study where exposures are known to the Investigator within the previous 4 months prior to admission to the clinic for this study or participated in a radiolabeled drug study where exposures are not known to the Investigator within the previous 6 months prior to admission to the clinic for this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2018-06-02 (Actual); Study Completion 2018-06-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics for napabucasin and metabolites by assessing plasma concentration | 1 week
Pharmacokinetics for napabucasin and metabolites by assessing urinary concentration | Up to 12 days
Pharmacokinetics for napabucasin and metabolites by assessing fecal concentration | Up to 12 days

SECONDARY OUTCOMES:
Number of Patients with Adverse Events | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States